CLINICAL TRIAL: NCT06456502
Title: Effectiveness of Non-invasive Neuromodulation Compared to Placebo on Sleep Quality in Patients With Post-COVID Symptoms: a Randomized Clinical Trial.
Brief Title: Effectiveness of Non-invasive Neuromodulation in Patients With Long-COVID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Stella María Fuensalida Novo, Proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 230220241322024
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Long-COVID; Post-acute COVID-19 Syndrome
Keywords: Post acute COVID-19 syndrome; Long-COVID; Non-invasive neuromodulation; Sleep quality; Depression; Anxiety; Fatigue; Quality of life; Pain
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders; Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: two armed parallel randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assignment to each group will be done by randomization software performed blindly by an external investigator who will not perform the interventions with the patients.
  Assessment will be performed by two persons of the team, not involved in the treatment.
  Participants will be blinded as they do not feel anything during the stimulation (whether within the active or placebo group), just the care provider will know if the cable is attached or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive neuromodulation (Experimental): The real treatment group using non-invasive neuromodulation
  Interventions: Device: Non-invasive neuromodulation
- PLACEBO (Placebo Comparator): The placebo treatment group (simulation of non-invasive neuromodulation application).
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Non-invasive neuromodulation — The treatment plan of non- invasive neuromodulation will be applied for two months, with a frequency of 2 weekly sessions of one hour duration, until completing a total of 15 sessions for each patient. The sessions will always be applied in the same time slot of the day (to avoid influence on the measurements, specially cortisol).
  Arms: Non-invasive neuromodulation
Other: Placebo — The treatment plan of placebo will be applied for two months, with a frequency of 2 weekly sessions of one hour duration, until completing a total of 15 sessions for each patient. Participants will be attached to the neuromodulation machine, however, the cable will not be connected. Participants will not be able to see the machine connections. The sessions will always be applied in the same time slot of the day (to avoid influence on the measurements, specially cortisol).
  Arms: PLACEBO

SUMMARY:
Sleep quality and duration are critical to cognitive, emotional and physical well-being, and poor sleep quality has been associated with an increased risk of cognitive, psychological and cardiometabolic disorders. Several important physiological activities occur during sleep including a reduction in heart rate and blood pressure. In addition, sleep exerts important modulatory effects on hormone release. Previous studies have shown that lack of sleep can generate exaggerated cortisol responses or psychological and physiological stressors. Cortisol has widespread effects throughout the body and brain, affecting mood, arousal, energy, metabolic processes, and immune and inflammatory system functioning. Therefore, disruptions in cortisol secretion during the night can influence a wide variety of processes in our body that may contribute to the perception of poorer sleep quality. In addition, the salivary enzyme α-amylase is considered a biomarker of cognitive, psychosocial, emotional or physical stress. It is important to note that the autonomic nervous system (ANS) regulates several physiological processes, including heart rate, blood pressure, respiration, and digestion. The ANS consists primarily of the sympathetic system and the parasympathetic system. Increased parasympathetic activity is considered to promote health, whereas a dominant or overactive sympathetic branch is considered to be detrimental to health.

A recent study found that both sleep quality and quantity of sleep were associated with resting ANS functioning. They found that poorer sleep quality was associated with greater sympathetic dominance. Research on the sympathetic and parasympathetic branches of the ANS has shown that autonomic imbalances are precursors to disease formation and other health-related risks. Coronavirus disease 2019 (COVID-19), has in many cases involved the presence of long-lasting symptoms several weeks or months after surviving acute infection with the virus, leading to a new disease called long COVID-19 or post-COVID-19 syndrome (PCS). A recent study showed that sleep quality influences the relationship between symptoms associated with sensitization and mood disorders with health-related quality of life in people suffering from long COVID.

Non-invasive neuromodulation directed to ANS may be an option to treat the sleep disorders observed in patients with long COVID.

OBJETIVES:

Therefore, the primary objective of this study is to evaluate the efficacy of a treatment protocol on the ANS by means of non-invasive neuromodulation in aspects related to sleep in long COVID patients compared to placebo. As secondary objectives, we propose to evaluate the efficacy of a treatment protocol on the ANS by non-invasive neuromodulation in aspects related to ANS functioning, psychological variables, fatigue, pain perception and quality of life in patients with long COVID.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with long COVID or post- acute COVID syndrome
* With a evolution of at least 6 months after acute SARS-cov-2 infection
* Whit symptoms present at baseline.

Exclusion Criteria:

* Pregnancy.
* Pacemakers
* Ulcerations or wounds in the area of electrode application.
* Decompensated heart disease.
* Epilepsy and/or choreic syndromes.
* Frequent medication with corticosteroids, hypnotics or supplements such as melatonin, Ashwagandha or phosphatidylserine.
* Hypersensitivity on hands and feet that influence the use of the gloves and socks from the neuromodulation system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Baseline, at the of 15th session, at 6 month an at one year
  The aspects of sleep to be assessed by means of the Pittsburgh sleep quality index (PSQI) scale and the sleep diary to be completed each morning and handed in on the last day of treatment.

SECONDARY OUTCOMES:
Heart variability | Baseline and at 8 weeks
  Through the We Cardio device, which provides variables such as resting heart rate (HRV) and the root mean square difference of successive interval between two successive R-waves (RMSSD), which reflects beat-to-beat variation in heart rate and is the main time-domain measure used to estimate vagal (parasympathetic) changes reflected in HRV.
Cortisol and alpha amylase levels | Baseline and at 8 weeks
  Cortisol and alpha amylase levels will be assessed with salivary tests that will be analyzed using a Soma cube reader device.
Psychological variables | Baseline, at 8 weeks, at 6 month an at one year
  Depression and anxiety will be evaluated by means of the hospital anxiety and depression scale (HADS) validated in spanish and with a high level of reliability and sensitivity for these variables
The quality of life | Baseline, at 8 weeks, at 6 month an at one year
  This variable will be evaluated by means of the EuroQol 5D (EQ-5D). It is a standardized instrument developed to describe and assess health-related quality of life (HRQoL)
Disability | Baseline, at 8 weeks, at 6 month an at one year
  The impact of the disease on patients will be assessed using the severe acute respiratory syndrome (SARS) functional impairment checklist (FIC), which is a questionnaire that assesses physical and psychological symptoms, as well as disability-related domains. The FIC has been shown to be valid, to show good reliability and to exhibit good psychometric properties for use as a tool to assess physical symptoms and disability-related domains in patients with SARS and patients with persistent COVID.
Pain intensity | Baseline, at 8 weeks, at 6 month an at one year
  Pain will be assessed by means of a numeric pain rating scale (NPRS), which allows measuring the intensity of pain described by the patient with maximum reproducibility between observers.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Fuensalida Novo, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Rey Juan Carlos University, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No